CLINICAL TRIAL: NCT03220373
Title: Predicting Early Treatment Termination (Dropout) and Post-treatment Clinical Outcome From Neuropsychological Functions in Abstinent Substance Use Dependent (SUD) Patients
Brief Title: Predicting Dropout and Outcome From Neuropsychological Functions in SUD Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Espen Walderhaug, Principal Investigator, Oslo University Hospital
Other Study IDs: 2015/11288
Record Dates: First submitted 2017-03-08; First posted 2017-07-18 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Substance Use Disorder (SUD)
Keywords: Neuropsychology; Cognition; Drop-out; Follow-up
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this project is to gain a more specific understanding of how different cognitive profiles predict residential treatment drop-out, treatment retention and post-treatment outcome in a population with Substance Use Disorder.

DETAILED DESCRIPTION:
This project collects the neuropsychological profile of residential SUD patients, in addition to treatment length, exit reason, hospital journal data and post-treatment clinical outcome data. The project aims to identify clinically relevant neurocognitive domains that predict treatment dropout and post-treatment clinical outcome. This will make it possible for future clinicians to focus their effort on neurocognitive functions most relevant for this particular patient group.

RESEARCH QUESTIONS:

1. What neurocognitive domain (and sub-domain) are the strongest predictor of treatment drop-out and retention?
2. What neurocognitive domain (and sub-domain) are the strongest predictor of post-treatment clinical outcome variables such as drug use, health and social integration.
3. Will data on treatment length, age, gender, substance abuse history or psychiatric co-morbidity predict outcome independently, or in interaction with, the neuropsychological profile?

This longitudinal prospective cohort study aims for a continuous collection of neuropsychological data baseline and post-treatment follow-up data until 2030.

ELIGIBILITY:
Inclusion Criteria:

* Substance Use Disorder (SUD) patients.
* 18 years or older.
* Qualified to consent to research participation.
* Able to speak and write in Norwegian.

Exclusion Criteria:

* Not qualified to consent to research participation.
* Insufficient understanding of Norwegian.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Treatment seeking Substance Use Disorder (SUD) patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-03-07 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Exit reason | On average 3 months
  Reason for terminating residential SUD treatment (Treatment completed or Drop-out)
Treatment retention | On average 3 months
  Number of days in treatment

SECONDARY OUTCOMES:
Substance use | 1 year after neuropsychological assessment
  DUDIT (Drug Use Disorders Identification Test)
Psychological distress | 1 year after neuropsychological assessment
  SCL-10 (Symptom Checklist)
Quality of Life | 1 year after neuropsychological assessment
  QoL-5 (Quality of Life)
ADHD symptoms | 1 year after neuropsychological assessment
  ASRS (ADHD Self-Report Scale)
Income | 1 year after neuropsychological assessment
  Nature of income
Housing | 1 year after neuropsychological assessment
  Nature of present accommodation

CONTACTS AND LOCATIONS:
Overall Officials: Espen Walderhaug, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway